CLINICAL TRIAL: NCT04221035
Title: High-Risk Neuroblastoma Study 2 of SIOP-Europa-Neuroblastoma (SIOPEN)
Acronym: HR-NBL2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001068-31; 2019/2894 (Other: CSET number (Gustave Roussy ID)); 2024-514917-36-00 (EU CTIS Number)
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: High-Risk Neuroblastoma; Patient With Insufficient Response Chemoimmunotherapy
MeSH Terms: interventions — Vincristine; Carboplatin; Etoposide; Vindesine; Dacarbazine; Ifosfamide; Doxorubicin; Busulfan; Melphalan; Thiotepa; Radiotherapy; dinutuximab; Cisplatin; Temozolomide; Irinotecan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- phase induction-R-I (Experimental): R-I: induction regimens RAPID COJEC vs GPOH Assuming a baseline 3-year EFS of 40%, with a sample size of 686 patients (343 in each arm) and a two-sided alpha=5% this trial will have 90% power to demonstrate an improvement of 12% in 3-year EFS, within a recruitment period of 3 years and a minimum follow up of 1.5 years.
  Patients with insufficient metastatic response at the end of induction chemotherapy, defined as SIOPEN score > 3 or less than 50% reduction in mIBG score (or > 3 bone lesions or less 50% reduction in number of FDG-PET-avid bone lesions for mIBG-non avid tumours), have a poorer prognosis.
  Chemoimmunotherapy arm Metastatic response rate after 4 courses of irinotecan-temozolomide (TEMIRI) combined with dinutuximab beta (DB) in patients with insufficient metastatic response at the end of induction chemotherapy (TEMIRI/DB).
  Interventions: Drug: Vincristine; Drug: Carboplatin; Drug: Etoposide; Drug: Vindesine; Drug: Dacarbazine; Drug: Ifosfamide; Drug: Doxorubicin; Drug: Dinutuximab Beta; Drug: Cisplatin; Drug: Temozolomide 100 MG; Drug: Irinotecan; Drug: Cyclophosphamid
- Phase high dose chemotherapy consolidation (Experimental): R-HDC: consolidation regimen Bu-Mel vs Thiotepa + Bu-Mel The 3-year EFS in the Bu-Mel arm (with immunotherapy) is estimated to be 55%. This study aims to show an improvement of 12% for the Thiotepa + Bu-Mel arm (3-year EFS of 67%). With a recruitment of 448 patients (224 in each arm) over a period of 3 years and a minimum follow-up of 2 years, the power to show a 12% difference is 80% (two-sided logrank test and α=5%).
  Interventions: Drug: Busulfan; Drug: Melphalan; Drug: Thiotepa
- Phase of radiotherapy (Experimental): R-RTx: 21.6 Gy radiotherapy vs 21.6 Gy + 14.4 Gy boost in patients with macroscopic residual disease
  Interventions: Radiation: Radiotherapy; Drug: Dinutuximab Beta

INTERVENTIONS:
Drug: Vincristine — 1.5 mg/m2 (max dose 2 mg)
  Other Names: L01CA02
  Arms: phase induction-R-I
Drug: Carboplatin — 750 mg/m2
  Other Names: LO1XA02
  Arms: phase induction-R-I
Drug: Etoposide — 175 mg/m2
  Other Names: L01CB01
  Arms: phase induction-R-I
Drug: Vindesine — 3 mg/m2/day (max dose 6 mg)
  Other Names: L01CA03
  Arms: phase induction-R-I
Drug: Dacarbazine — 200 mg/m2/day
  Other Names: L01AX04
  Arms: phase induction-R-I
Drug: Ifosfamide — 1500 mg/m2/day
  Arms: phase induction-R-I
Drug: Doxorubicin — 30 mg/m2/dose
  Other Names: L01DB01
  Arms: phase induction-R-I
Drug: Busulfan — < 9kg: 1.0 mg/kg/dose 9 kg to < 16 kg : 1.2 mg/kg/dose 16 kg to 23 kg : 1.1 mg/kg/dose >23 kg to 34 kg: 0.95 mg/kg/dose >34 kg: 0.8 mg/kg/dose Infusion IV over 2 hours Administration every 6 hours for a total of 16 doses
  Other Names: L01AB01
  Arms: Phase high dose chemotherapy consolidation
Drug: Melphalan — 140 mg/m2/dose IV short infusion (15'), at least 24 h after the last busulfan dose
  Other Names: L01AA03
  Arms: Phase high dose chemotherapy consolidation
Drug: Thiotepa — 300 mg/m2/day over 2 hours
  Other Names: L01AC01
  Arms: Phase high dose chemotherapy consolidation
Radiation: Radiotherapy — 21.6 Gy 21.6 Gy + boost de 14.4 Gy
  Arms: Phase of radiotherapy
Drug: Dinutuximab Beta — Patients >12 kg are dosed based on the BSA: 10 mg/m^2/day Patients ≤ 12 kg are dosed according to their body weight: 0.33 mg/kg/day
  Other Names: L01XC16
  Arms: Phase of radiotherapy; phase induction-R-I
Drug: Cisplatin — 80 mg/m2/24h
  Other Names: L01XA01
  Arms: phase induction-R-I
Drug: Temozolomide 100 MG — 100 mg/m²/Day
  Arms: phase induction-R-I
Drug: Irinotecan — 50 mg/m²/jour de J0 à J4
  Arms: phase induction-R-I
Drug: Cyclophosphamid — Cyclophosphamide has been demonstrated to have a cytostatic effect in many tumour types. The active metabolites of cyclophosphamide are alkylating agents which transfer alkyl groups to DNA during the process of cell division, thus preventing normal synthesis of DNA.
  Arms: phase induction-R-I

SUMMARY:
This is an international multicenter, open-label, randomized phase III trial including three sequential randomizations to assess efficacy of induction and consolidation chemotherapies and radiotherapy for patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
This is an international multicenter, open-label, randomized phase III trial including three sequential randomizations to assess efficacy of induction and consolidation chemotherapies and radiotherapy for patients with high-risk neuroblastoma.

The first randomization (R-I) will compare the efficacy of two induction chemotherapies (RAPID COJEC and GPOH regimens) in a phase III setting. The primary endpoint will be the 3-year EFS from date of randomization . The R-I randomization will be stratified on age, stage, MYCN status and countries.

The second randomization (R-HDC) will compare the efficacy of single HDC with Bu-Mel versus tandem HDC with Thiotepa followed by Bu-Mel. The primary endpoint is 3-year EFS calculated from the date of the R-HDC randomization. The R-HDC randomization will be stratified on the age, stage, MYCN status, induction chemotherapy regimen, response to induction phase and countries.

The impact of local treatment in this phase III setting will be assessed, according to the presence or not of a macroscopic residual disease after surgery and HDC.

In case of macroscopic residual disease, 21.6 Gy radiotherapy to the preoperative tumor bed will be randomized (R-RTx) versus the same treatment plus a sequential boost of additional 14.4 Gy to the residual tumor. The primary endpoint of R-RTx is 3-year EFS from the date of the R-RTx randomization. The R-RTx randomization will be stratified on age, stage, MYCN status, induction chemotherapy regimen, HDC regimen and countries.

In case of no macroscopic residual disease, 21.6 Gy radiotherapy will be delivered to the preoperative tumor bed.

ELIGIBILITY:
Inclusion Criteria:

Enrollment in HR-NBL2 will be performed:

* at diagnosis before the beginning of chemotherapy or
* up to 21 days after one course of Carboplatin-Etoposide for patients with localized neuroblastoma or infants with metastatic neuroblastoma with MYCN amplification or patients with metastatic neuroblastoma treated in emergency or
* up to 21 days after one course of the current protocol for R-I randomisation (RAPID COJEC/GPOH) low/intermediate risk neuroblastoma in Germany/Netherlands for patients with localized neuroblastoma or infants with metastatic neuroblastoma with MYCN amplification

HR-NBL2 eligibility criteria:

1. Established diagnosis of neuroblastoma according to the SIOPEN- modified International Neuroblastoma Risk Group (INRG) criteria, High-risk neuroblastoma defined as:

   * Stage M neuroblastoma above 365 days of age at diagnosis (no upper age limit) and Ms neuroblastoma 12-18 months old, any MYCN status or
   * L2, M or Ms neuroblastoma any age with MYCN amplification, or focal high level MYC or MYCL amplification.

   In Germany, patients aged less than 18 months with stage M and without MYCN amplification will not be enrolled in HR-NBL2 trial.
2. No previous chemotherapy or up to 21 days after one cycle of Carboplatin-Etoposide chemotherapy for patients with localized neuroblastoma or infants with metastatic neuroblastoma with MYCN amplification or patients with metastatic neuroblastoma treated in emergency or up to 21 days after one course of the current protocol for low/intermediate risk neuroblastoma in Germany/Netherlands for patients with localized neuroblastoma or infants with metastatic neuroblastoma with MYCN amplification
3. Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to initiation of treatment. Sexually active patients must agree to use acceptable and appropriate contraception while on HR-NBL2 study and for one year after stopping the study. Acceptable contraception is defined in CTFG Guidelines "Recommendations related to contraception and pregnancy testing in clinical trials" (Appendix 11). Female patients who are lactating must agree to stop breast-feeding.
4. Written informed consent to enter the HR-NBL2 protocol from patient or parents/legal representative, patient, and age-appropriate assent.
5. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.
6. Patients should be able and willing to comply with study visits and procedures as per protocol

R-I eligibility criteria:

- Written informed consent to enter the R-I randomisation from patient or parents/legal representative, patient, and age- appropriate assent.

In case of parents'/patient's refusal to R-I, or Organ toxicity exclusion criteria at diagnosis, patients can still be enrolled in HR- NBL2 trial with parents'/patient's consent before or within 3 weeks from the beginning of chemotherapy

R-HDC randomisation (Single HDC Bu-Mel/ Tandem HDC Thiotepa+Bu-Mel) Etoposide or one course of the current protocol for low/intermediate risk neuroblastoma in Germany/Netherlands). Patients will be treated with the standard induction regimen per country (Rapid COJEC or GPOH) and will be potentially eligible for subsequent randomisations.

Randomisation for HDC strategy will be performed at the end of induction after the disease evaluation and after surgery of the primary tumour for those patients who will receive surgery before HDC.

R-HDC eligibility criteria:

1. - Stage M neuroblastoma above 365 days of age at diagnosis, any MYCN status, EXCEPT patients with stage M or Ms 12-18 months old with numerical chromosomal alterations only, and in complete metastatic response at the end of induction: in this case, patients will have surgery and no further treatment.

   OR

   - L2, M or Ms neuroblastoma, any age, with MYCN amplification, or focal high level MYC or MYCL amplification
2. Age < 21 years at the time of randomization
3. Complete response (CR) or partial response (PR) at metastatic sites:

   * Bone disease: mIBG uptake completely resolved or SIOPEN score ≤ 3 and at least 50% reduction in mIBG score (or ≤ 3 bone lesions and at least 50% reduction in number of FDG- PET-avid bone lesions for mIBG-nonavid tumours).
   * Bone marrow disease: CR and/or minimal disease (MD) according to International Neuroblastoma Response Criteria
   * Other metastatic sites: CR. (after induction chemotherapy +/- surgery), except for distant lymph nodes for which PR is accepted with a possible secondary surgery
4. Acceptable organ function and performance status:

   * Performance status ≥ 50%.
   * Hematological status: ANC>0.5x109/L, platelets > 20x 109/L
   * Cardiac function: (< grade 2)
   * Normal chest X-Ray and oxygen saturation.
   * Absence of any toxicity ≥ grade 3. 4) Sufficient collected stem cells available; a total harvest of at least 6 x 106/kg CD34+ cells, to be stored in at least 4 separate bags to administer at least 3 x 106/kg CD34+ cells per rescue.
5. Written informed consent, including agreement of patient or parents/legal guardian for minors, to enter the R-HDC randomisation.
6. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.
7. Patients should be able and willing to comply with study visits and procedures as per protocol.

In case of parents'/patient's refusal, or insufficient stem cells, collection for tandem HDC but with a minimum of 3 x 106 CD34+ cells/kg body weight, or in case of patients older than 21 years, or organ toxicity, HDC will consist on the standard HD Bu-Mel and patients will be eligible for the subsequent randomisation.

R-RTx randomisation (Local Radiotherapy) Chemoimmunotherapy arm

R-RTx eligibility criteria:

An evaluation of the local disease will be performed after HDC/ASCR and surgery:

* In case of no local macroscopic disease, all patients will receive 21,6-Gy radiotherapy to the pre-operative tumour bed
* In case of local macroscopic residual disease, patients will be eligible to R-RTx if the following criteria are met:

  1. No evidence of disease progression after HDC/ASCR.
  2. Interval between the last ASCR and radiotherapy start between 60 and 90 days.
  3. Performance status greater or equal 50%.
  4. Hematological status: ANC >0.5x109/L, platelets > 20x109/L.
  5. Written informed consent, including agreement of patient or parents/legal guardian for minors, to enter the R-RTx randomisation.
  6. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.
  7. Patients should be able and willing to comply with study visits and procedures as per protocol.

In case of parents'/patient's refusal of the randomisation, the patient will receive 21.6 Gy radiotherapy to the pre-operative tumour bed.

Chemoimmunotherapy arm eligibility criteria:

1. Insufficient metastatic response at the end of induction chemotherapy, defined as:

   * SIOPEN score > 3 or less than 50% reduction in mIBG score (or > 3 bone lesions or less 50% reduction in number of FDG-PET-avid bone lesions for mIBG-non avid tumours) OR
   * Bone marrow disease: SD according to International Neuroblastoma Response Criteria OR
   * Other metastatic sites: PR or SD. For distant lymph nodes: PR and not resectable or SD.
2. Performance status ≥ 50%.
3. Hematological status: ANC>0.75x109/L without G-CSF for at least 48 hours (or ANC ≥ 0.50 x 109 /L in case of bone marrow involvement), platelets > 50x 109/L and rising, without platelets transfusion for 72 hours.
4. AST or ALT ≤7.5 ULN and total bilirubin ≤1.5 ULN. In patients with liver metastases, total bilirubin ≤2.5 ULN is allowed.
5. No active infection;
6. No grade >2 gastrointestinal toxicity.
7. No grade ≥ 3 toxicity related to previous treatment.
8. Oxygen saturation > 94%

Non-inclusion criteria for HR-NBL2:

1. Any negative answer concerning the HR-NLB2 inclusion criteria
2. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving his consent.
3. Participating in another clinical study with an IMP while on study treatment.
4. Chronic inflammatory bowel disease and/or bowel obstruction.
5. Pregnant or breastfeeding women.
6. Known hypersensitivity to the active substance or to any of the excipients of the study drugs
7. Concomitant self-medication medicine that in the investigator opinion could interact with study treatments, including herbal medicine (e.g. St John's Wort (Hypericum Perforatum).

Non-inclusion criteria specific to the R-I randomisation (RAPID COJEC/GPOH):

1. Urinary tract obstruction ≥ grade 3
2. Heart failure or myocarditis ≥ grade 2, any arrhythmia or myocardial infection
3. Peripheral motor or sensory neuropathy ≥ grade 3
4. Demyelinating form of Charcot-Marie-Tooth syndrome
5. Hearing impairment ≥ grade 2
6. Concurrent prophylactic use of phenytoin
7. Cardiorespiratory disease that contraindicates hyperhydration

Non-inclusion criteria common to all randomisations (R-I, R-HDC, and R-RTx):

1. Any negative answer concerning the inclusion criteria of R-I or R- HDC or R-RTx will render the patient ineligible for the corresponding therapy phase randomisation. However, these patients may remain on study and be considered to receive standard treatment of the respective therapy phase, and may be potentially eligible for subsequent randomisations.
2. Liver function: Alanine aminotransferase (ALT) > 3.0 x ULN and blood bilirubin > 1.5 x ULN (toxicity ≥ grade 2). In case of toxicity ≥ grade 2, call national principal investigator study coordinator to discuss the feasibility.
3. Renal function: Creatinine clearance and/or GFR < 60 ml/min/1.73m² (toxicity ≥ grade 2). If GFR < 60ml/min/1.73m², call national principal investigator study coordinator to discuss about the treatment.
4. Dyspnea at rest and/or pulse oximetry <95% in air (only for R-HDC, and R-RTx)
5. Any uncontrolled intercurrent illness or infection that in the investigator opinion would impair study participation.
6. Concomitant use with yellow fever vaccine and with live virus or bacterial vaccines.
7. Patient allergic to peanut or soya.

Non-inclusion criteria to R-HDC:

- Any negative answer concerning the R-HDC inclusion criteria

Non-inclusion criteria to chemoimmunotherapy arm:

- Any negative answer concerning the inclusion criteria of chemoimmunotherapy arm.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | Assessed at each end of randomization sequences up to one year
  Event free survival

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Pasqualini, MD PhD, Study Chair — Gustave roussy, Paris, France
Locations (142):
- Australia (7):
  - Sydney children Hospital, Sydney, Randwick
  - Children's Cancer Centre, Monash Children's Hospital, Clayton
  - Oncology/Haematology Department, Perth Children's Hospital, Nedlands
  - Children's Cancer & Haematology Services, John Hunter Children's Hospital, New Lambton Heights
  - Australian and New Zealand Children's Hematology/oncology Group, Sydney
  - sydney children Hospital, Sydney
  - Cancer Centre for Children, The Children's Hospital, Westmead
- Austria (5):
  - Medical University Graz, Graz
  - Landeskrankenhaus-Universitätsklinikum Innsbruck, Innsbruck
  - Kepler Universitatsklinikum Linz, Linz
  - Universitastsklinikum Salzburg, Salzburg
  - St Anna'S Children Hospital, Vienna
- Belgium (5):
  - Hôpital Universitaire des Enfants Reine Fabiola (ULB), Brussels
  - Cliniques Universitaires Saint-Luc (UCL), Brussels
  - University Hospital Gent, Ghent
  - University Hospitals Leuven, Leuven
  - CHR Citadelle, Liège
- Czechia (2):
  - University Hospital Motol, Prague, Prague
  - Klinika dětské onkologie FN Brno, Brno
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Department of Paediatrics and Adolescent Medicine, Rigshospitalet, Copenhagen
  - The Hans Christian Andersen Children's Hospital, University of Southern Denmark, Odense
- Finland (5):
  - New Children's Hospital, Helsinki University Hospital, Helsinki and Uusimaa Hospital District, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (37):
  - Gustave Roussy, Villejuif, Val De Marne
  - CHU d'AMIENS, Amiens
  - CHU angers, Angers
  - CHU-Pôle Médico-Chirurgical de l'Enfant et l'Adolescant, Besançon
  - CHU Bordeaux, Bordeaux
  - Groupe Hospitalier Pellegrin - Chu - Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Brest - Hôpital du Morvan, Brest
  - Centre François Baclesse, Caen
  - CHU de Caen, Caen
  - CHU Estaing, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Hopital d'enfants Marechal de lattre, Dijon
  - Hôpital Couple-Enfant CHU de Grenoble, Grenoble
  - Chu de La Reunion - St Denis, La Réunion
  - centre Oscar lambert, Lille
  - Hôpital de la Mère et de l'Enfant - CHU Limoges, Limoges
  - Centre Léon Berard, Lyon
  - hopital la Timone, Marseille
  - CHRU Nancy-Hôpital Brabois Enfant, Nancy
  - Institut de cancérologie de Loraine, Nancy
  - Centre Antoine Lacassagne, Nice
  - CHU Nice-Hôpital d'Archet, Nice
  - Hôpital Armand Trousseau, Paris
  - institut Curie, Paris
  - CHU Poitiers, Poitiers
  - Hôpital Américain -CHU Reims, Reims
  - Centre Eugène Marquis, Rennes
  - CHU Rennes, Rennes
  - Hôpital des Enfants - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - Institut de cancérologie de l'Ouest - Sité René Gauducheau, Saint-Herblain
  - CHU Haute Pierre, Strasbourg
  - Institut de Cancérologie Strasbourg, Strasbourg
  - Hopital des enfants-CHU Toulouse, Toulouse
  - IUCT Oncopole, Toulouse
  - CHU Tours Hôpital Clocheville, Tours
- Germany (2):
  - charite universitatsmedizin Berlin, Berlin
  - Uniklinik Köln, Klinik und Poliklinik für Kinder und Jugendmedizin, Cologne
- Greece (7):
  - Children's General Hospital "I AGHIA SOFIA", Athens
  - Children's General Hospital "P. & A. KYRIAKOU", Athens
  - "MITERA" Private, General, Obstetrics - Gynaecology, Paediatric Clinic S.A., Athens
  - Children's General Hospital "AGHIA SOFIA", Athens
  - University General Hospital of Heraklion (UnGHH), Heraklion
  - University General Hospital of Thessaloniki "AHEPA", Thessaloniki
  - General Hospital of Thessaloniki "IPPOKRATIO", Thessaloniki
- RAMBAM Medical Center, Haifa, Israel
- Italy (12):
  - A.O.U Policlinico di Bari, Bari
  - Spedali civili Ospedale Dei Bambini Oncoematologia pediatrica e TMO, Brescia
  - policlinico rodolico San marco, Catania
  - Azienda ospedaliero universtaria Anna Meyer, Florence
  - instituto Giannina Gaslini genova, Genova
  - IRCCS "Istituto Giannina Gaslini", Genova
  - Azienda Policlinico di Modena, Modena
  - Azienda ospedaliero universitaria di Parma, Parma
  - Policlino San matteo di Pavia, Pavia
  - U.O Pediatria, SS Oncoematologia pediatrica, Rimini
  - IRCCS Burlo Garoflo oncoematologia, Trieste
  - U.O.C oncoematologia pediatrica ospedale Donna Bambino, Verona
- Lithuania (2):
  - Vilnius University Hospital Santaros Klinikos, Vilnius
  - National Cancer Institute, Vilnius
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Princess Maxima center, Utrecht
- Norway (4):
  - Haukeland University Hospital, Haukeland
  - Oslo University Hospital, Oslo
  - University Hospital Northern Norway, Tromsoe, Tromsø
  - St Olavs Hospital,, Trondheim
- Slovakia (3):
  - Children's University Hospital Banská Bystrica, Banská Bystrica
  - NÚDCH- National Institute of Children's Diseases,, Bratislava
  - Children's University Hospital Košice, Košice
- University medical center Ljubljana, University Children's Hospital Ljubljana, Slovenia, Ljubljana, Slovenia
- Spain (11):
  - Hospital Universitario Son Espases, Balea
  - Hospital Universitario Vall D´Hebron, Barcelona
  - Hospital Universitario Cruces, Cruces
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario Infantil Niño Jesús, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Politécnico de La FE, Valencia
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm, Stockholm
  - Norrland University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (9):
  - Kantonsspital Aarau AG Klinik für Kinder und Jugendliche, Aarau
  - Universitäts-Kinderspital beider Basel (UKBB), Basel
  - Ospedale San Giovanni Pediatria, Emato-oncologia pediatrica, Bellinzona
  - Inselspital, Universitätsklinik für Kinderheilkunde, Bern
  - HUG Hôpitaux Universitaires de Genève Unité d'Hémato-Oncologie Pédiatrique, Geneva
  - CHUV - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonsspital, Kinderspital pädiatrische Hämatologie/Onkologie, Lucerne
  - Ostschweizer Kinderspital Hämatologie/Onkologie Claudiusstrasse 6, Sankt Gallen
  - Division of Pediatric Oncology Universitäts-Kinderspital Zürich, Zurich
- United Kingdom (18):
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham children's Hospital, Birmingham
  - University Hospitals Birmingham Queen Elisabeth Hospital(UHB), Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Addenbrookes Hospital, Cambridge, Cambridge
  - Noah's Ark Children's Hospital for Wales - Cardiff, Cardiff
  - Royal Hospital for Sick Children - Edinburgh, Edinburgh
  - Royal Hospital for Children Glasgow, Glasgow
  - Leeds General Infirmary, Leeds
  - Alder Hey Children's Hospital - Liverpool, Liverpool
  - Great Ormond Street Hospital - London, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle, Newcastle
  - Nottingham Children's Hospital, Nottingham
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR